CLINICAL TRIAL: NCT02289963
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Alirocumab in High Cardiovascular Risk Patients With Hypercholesterolemia Not Adequately Controlled With Their Lipid-Modifying Therapy in South Korea and Taiwan
Brief Title: Evaluation of Alirocumab in Addition to Lipid-Modifying Therapy in Patients With High Cardiovascular Risk and Hypercholesterolemia in South Korea and Taiwan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC14074; U1111-1157-3294 (Other: UTN)
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: Yes

ARMS (2):
- Placebo Q2W (Placebo Comparator): Placebo (for alirocumab) subcutaneous (SC) injection every 2 weeks (Q2W) added to stable Lipid-Modifying Therapy (LMT) for 24 weeks.
  Interventions: Drug: Placebo (for Alirocumab); Drug: Lipid-Modifying Therapy (LMT)
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W (Placebo Comparator): Alirocumab 75 mg SC injection Q2W added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) at Week 8.
  Interventions: Drug: Alirocumab; Drug: Lipid-Modifying Therapy (LMT)

INTERVENTIONS:
Drug: Placebo (for Alirocumab) — Solution for injection, one subcutaneous injection in the abdomen with a disposable auto-injector.
  Arms: Placebo Q2W
Drug: Alirocumab — Solution for injection, one subcutaneous injection in the abdomen with a disposable auto-injector.
  Other Names: SAR236553; REGN727; Praluent®
  Arms: Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Drug: Lipid-Modifying Therapy (LMT) — Statins (Rosuvastatin, Simvastatin or Atorvastatin) at stable dose with or without other LMT as clinically indicated.

SUMMARY:
Primary Objective:

To demonstrate the reduction of low-density lipoprotein cholesterol (LDL-C) by alirocumab as add-on therapy to stable maximally tolerated daily statin therapy with or without other lipid-modifying therapy (LMT) in comparison with placebo after 24 weeks of treatment in high cardiovascular risk participants with hypercholesterolemia in South Korea and Taiwan.

Secondary Objectives:

* To evaluate the effect of alirocumab in comparison with placebo on LDL-C after 12 weeks of treatment.
* To evaluate the effect of alirocumab on other lipid parameters: apolipoprotein B (Apo B), non high-density lipoprotein cholesterol (non-HDL-C), total cholesterol (TC), lipoprotein (a) (Lp [a]), high-density lipoprotein cholesterol (HDL-C), triglycerides (TGs), and apolipoprotein A-1 (Apo A-1).
* To evaluate the safety and tolerability of alirocumab.
* To evaluate the development of anti-alirocumab antibodies (ADA).

DETAILED DESCRIPTION:
The maximum study duration was approximately 35 weeks per participant, including up to 3 weeks screening period, 24 weeks double-blind treatment period, and 8 weeks follow-up period.

ELIGIBILITY:
Inclusion criteria:

Participants with hypercholesterolemia and established coronary heart disease (CHD) or CHD risk equivalents who are not adequately controlled with a maximally tolerated daily dose of statin with or without other LMT, both at stable dose for at least 4 weeks prior to screening visit (Week -3).

Exclusion criteria:

* Aged <18 years or legal age of adulthood, whichever was greater.
* Participants without established CHD or CHD risk equivalent.
* LDL-C <70 mg/dL (<1.81 mmol/L) in participants with a history of documented cardiovascular disease.
* LDL-C <100 mg/dL (<2.59 mmol/L) in participants without a history of documented cardiovascular disease.
* Not on a stable dose of LMT (including statin) for at least 4 weeks prior to the screening visit (Week -3) or between screening to randomization visits.
* Currently taking a statin other than atorvastatin, rosuvastatin or simvastatin.
* Atorvastatin, rosuvastatin or simvastatin was not taken daily or not taken at a registered dose.
* Daily doses above atorvastatin 80 mg, rosuvastatin 20 mg or simvastatin 40 mg.
* Fasting serum triglycerides >400 mg/dL (>4.52 mmol/L) at the screening period.

The above information is not intended to contain all considerations relevant to a participants's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (27):
- South Korea (16):
  - Investigational Site Number 410001, Anyang
  - Investigational Site Number 410009, Anyang-si
  - Investigational Site Number 410017, Busan
  - Investigational Site Number 410007, Busan
  - Investigational Site Number 410002, Daegu
  - Investigational Site Number 410011, Goyang-si
  - Investigational Site Number 410003, Gwangju
  - Investigational Site Number 410012, Incheon
  - Investigational Site Number 410018, Jeonju
  - Investigational Site Number 410006, Seoul
  - Investigational Site Number 410004, Seoul
  - Investigational Site Number 410015, Seoul
  - Investigational Site Number 410008, Seoul
  - Investigational Site Number 410005, Seoul
  - Investigational Site Number 410010, Seoul
  - Investigational Site Number 410013, Ulsan
- Taiwan (11):
  - Investigational Site Number 158007, Changhua
  - Investigational Site Number 158005, Hsinchu
  - Investigational Site Number 158011, Kaohsiung City
  - Investigational Site Number 158010, Kaohsiung City
  - Investigational Site Number 158006, Taichung
  - Investigational Site Number 158008, Tainan
  - Investigational Site Number 158009, Tainan Hsien
  - Investigational Site Number 158001, Taipei
  - Investigational Site Number 158003, Taipei
  - Investigational Site Number 158002, Taipei
  - Investigational Site Number 158004, Taoyuan Hsien

REFERENCES:
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- [Derived] Chao TH, Hsiao PJ, Liu ME, Wu CJ, Chiang FT, Chen ZC, Chen CP, Yeh HI, Lee TH, Chiang CE. A subanalysis of Taiwanese patients from ODYSSEY South Korea and Taiwan study evaluating the efficacy and safety of alirocumab. J Chin Med Assoc. 2019 Apr;82(4):265-271. doi: 10.1097/JCMA.0000000000000062. PMID 30946207
- [Derived] Koh KK, Nam CW, Chao TH, Liu ME, Wu CJ, Kim DS, Kim CJ, Li I, Li J, Baccara-Dinet MT, Hsiao PJ, Chiang CE. A randomized trial evaluating the efficacy and safety of alirocumab in South Korea and Taiwan (ODYSSEY KT). J Clin Lipidol. 2018 Jan-Feb;12(1):162-172.e6. doi: 10.1016/j.jacl.2017.09.007. Epub 2017 Oct 19. PMID 29153823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 27 centers in South Korea and Taiwan. Overall 316 participants were screened between January and September 2015, of whom 117 were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Randomization was stratified according to prior history of myocardial infarction (MI) or ischemic stroke, intensity of statin treatment and country. Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 1:1 ratio (Placebo:Alirocumab). A total of 199 participants were randomized.
Groups:
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W: Alirocumab 75 mg SC injection Q2W added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when low-density lipoprotein cholesterol (LDL-C) levels ≥70 mg/dL (1.81 mmol/L) at Week 8.
Period: Overall Study
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Started | 102 (Randomized) | 97 (Randomized)
Treated | 102 | 97
Completed | 97 | 87
Not Completed | 5 | 10
Not completed — Adverse Event | 1 | 2
Not completed — Poor compliance to protocol | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Last injection missed | 2 | 2
Not completed — End treatment visit outside visit window | 0 | 4
Not completed — Other than specified above | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Placebo Q2W: Placebo (for alirocumab) SC injection Q2W added to stable LMT for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Total
Number analyzed (Participants) | 102 | 97 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (9.1) | 61.2 (10.4) | 60.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 14 | 35
  Male | 81 | 83 | 164
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] — Calculated LDL-C in mmol/L from Friedewald formula (LDL-C = Total cholesterol - High-density lipoprotein cholesterol [HDL-C] - [Triglyceride/2.2]).
  mmol/L | 2.572 (0.653) | 2.513 (0.721) | 2.543 (0.686)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent-to-Treat (ITT) Analysis
Description: Adjusted Least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data up to Week 24 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 24
Population: ITT population that included all randomized participants with one baseline and at least one post-baseline calculated LDL-C on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percent change | 6.3 (2.9) | -57.1 (3.0)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; Alirocumab group was compared to placebo group using an appropriate contrast statement; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; Least Square (LS) Mean Difference = -63.4, 95% CI 2-sided [-71.6 to -55.2] — Alirocumab 75 mg Q2W/ Up to 150 mg Q2W vs. Placebo Q2W

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data up to Week 24 (i.e. up to 21 days after last injection) (on-treatment analysis).
Time Frame: From Baseline to Week 24
Population: Modified ITT (mITT) population that included all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 100 | 97
Percent Change | 6.0 (2.7) | -60.2 (2.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance was at 0.05 level; LS Mean Difference = -66.2, 95% CI 2-sided [-73.9 to -58.4] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 were obtained from MMRM model including all available post-baseline data up to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percent change | 4.7 (2.2) | -57.9 (2.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -62.5, 95% CI 2-sided [-68.8 to -56.3] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 were obtained from MMRM model including available post-baseline on-treatment data up to Week 24 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 24
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 100 | 97
percent change | 4.7 (2.2) | -58.4 (2.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -63.1, 95% CI 2-sided [-69.2 to -57.0] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including all available post-baseline data up to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment (Apo B ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 100 | 96
percent change | 4.1 (2.3) | -42.3 (2.4)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -46.3, 95% CI 2-sided [-53.0 to -39.7] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

6. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 - On-treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data up to Week 24 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 24
Population: Participants of the mITT population with one baseline and at least one post-baseline Apo B value on-treatment (Apo B mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 99 | 95
percent change | 3.8 (2.1) | -45.4 (2.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -49.2, 95% CI 2-sided [-55.3 to -43.1] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

7. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment (non-HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percent change | 4.3 (2.4) | -47.2 (2.5)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -51.5, 95% CI 2-sided [-58.4 to -44.6] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 - On-treatment Analysis
Description: as for outcome 6
Time Frame: From Baseline to Week 24
Population: Participants of the mITT population with one baseline and at least one post-baseline non-HDL-C value on-treatment (non-HDL-C mITT population).
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 100 | 97
percent change | 4.1 (2.2) | -50.1 (2.3)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -54.2, 95% CI 2-sided [-60.6 to -47.8] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Total-C value on- or off-treatment (Total-C ITT population).
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percent change | 4.0 (1.8) | -31.2 (1.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -35.2, 95% CI 2-sided [-40.3 to -30.1] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

10. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: Apo B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 100 | 96
percent change | 5.2 (1.8) | -40.9 (1.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -46.1, 95% CI 2-sided [-51.2 to -41.0] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

11. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: Non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percent change | 3.9 (1.8) | -47.3 (1.9)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -51.2, 95% CI 2-sided [-56.4 to -46.1] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

12. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: Total-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percent change | 2.8 (1.4) | -32.9 (1.4)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -35.8, 95% CI 2-sided [-39.7 to -31.9] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

13. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 were obtained from multiple imputation approach model for handling of missing data. All available post-baseline data up to Week 24 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percentage of participants | 14.2 | 85.8
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 46.9, 95% CI 2-sided [18.4 to 119.4] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

14. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - On-treatment Analysis
Description: Adjusted percentages at Week 24 were obtained from multiple imputation approach model including available post-baseline on-treatment data up to Week 24 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 100 | 97
percentage of participants | 14.1 | 88.8
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 70.0, 95% CI 2-sided [23.3 to 210.8] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

15. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 were obtained from multiple imputation approach followed by robust regression model for handling of missing data. All available post-baseline data up to Week 24 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percent change | -2.251 (2.962) | -35.862 (3.011)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Robust — Threshold for significance at 0.05 level; Multiple imputation approach followed by a robust regression model; Adjusted Mean Difference = -33.611, 95% CI 2-sided [-41.883 to -25.338] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

16. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein (HDL-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment (HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percent change | 6.2 (1.7) | 13.8 (1.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0029, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = 7.5, 95% CI 2-sided [2.6 to 12.4] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

17. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 were obtained from multiple imputation approach followed by robust regression model including all available post-baseline data up to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percent change | -3.627 (3.111) | -8.143 (3.204)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg Q2W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.3110, Regression, Robust — Threshold for significance at 0.05 level; Multiple imputation approach followed by a robust regression model; LS Mean Difference = -4.515, 95% CI 2-sided [-13.250 to 4.219] — Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs. Placebo Q2W

18. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 (Apo A-1) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo A-1 value on- or off-treatment (Apo A-1 ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 100 | 96
percent change | 3.2 (1.2) | 4.5 (1.2)

19. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 12- ITT Analysis
Description: Adjusted means and standard errors at Week 12 were obtained from multiple imputation approach followed by robust regression model including all available post-baseline data up to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percent change | -1.676 (2.732) | -33.601 (2.778)

20. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percent change | 2.0 (1.5) | 7.1 (1.6)

21. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 were obtained from multiple imputation approach followed by a robust regression model including all available post-baseline data up to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 102 | 97
percent change | 2.113 (3.192) | -6.999 (3.252)

22. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: Apo A-1 ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Number analyzed (Participants) | 100 | 96
percent change | 1.5 (1.1) | 4.5 (1.1)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 32 post-treatment follow-up visit) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'treatment emergent period' (the time from the first dose of study drug up to the last dose of study drug +70 days).
Groups:
- Placebo Q2W: Participants exposed to Placebo (for Alirocumab) SC injection Q2W added to stable LMT (mean exposure of 23 weeks).
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W: Participants exposed to Alirocumab 75 mg Q2W/up to 150 mg Q2W SC injection added to stable LMT (mean exposure of 24 weeks).
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/102 | 1/97
Serious Adverse Events (participants affected / at risk) | 10/102 | 17/97
Other Adverse Events (participants affected / at risk) | 15/102 | 19/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=102) | Alirocumab 75 mg Q2W/Up to 150 mg Q2W (N=97)
Influenza (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cervical myelopathy (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Neuromuscular pain (Nervous system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Brachiocephalic artery stenosis (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Loss of anatomical alignment after fracture reduction (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Device failure (Product Issues) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=102) | Alirocumab 75 mg Q2W/Up to 150 mg Q2W (N=97)
Nasopharyngitis (Infections and infestations) | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 6 | 3
Dizziness (Nervous system disorders) | 3 | 6
Headache (Nervous system disorders) | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.